CLINICAL TRIAL: NCT07032337
Title: Efficacy and Safety of Conventional Immunosuppressant Therapies in Elderly Patients With Neuromyelitis Optica Spectrum Disorder: A Target Trial Emulation Study
Brief Title: Efficacy and Safety of Conventional Immunosuppressant Therapies in Elderly Patients With Neuromyelitis Optica Spectrum Disorder
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Ju-Hong Min, Professor, Samsung Medical Center
Other Study IDs: IST_NMOSD
Record Dates: First submitted 2025-04-24; First posted 2025-06-23 (Actual); Last update posted 2025-06-23 (Actual); Status verified 2025-06

CONDITIONS: Neuromyelitis Optica Spectrum Disorder (NMOSD)
Keywords: immunosuppressive therapies; azathioprine; mycophenolate mofetil; rituximab; elderly
MeSH Terms: conditions — Neuromyelitis Optica

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IST group: patients who initiated any ISTs
- non-IST group: patients who did not initiate any ISTs

SUMMARY:
Newly diagnosed NMOSD patients

DETAILED DESCRIPTION:
From 2011 to 2022, newly diagnosed NMOSD patients who had not previously claimed NMOSD. Exclusion criteria were history of cancer or had used ISTs (excluding steroids) prior to the NMOSD diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* From 2011 to 2022, newly diagnosed NMOSD patients..

Exclusion Criteria:

* Patients had a history of cancer
* Patients had used ISTs (excluding steroids) prior to the NMOSD diagnosis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Once diagnosed, patients were eligible to enter weekly emulated trials starting from the diagnosis date. At the beginning of each week (baseline of each emulated trial), eligibility was reassessed: patients who developed cancer or had previously initiated ISTs been excluded from the trial. Eligible patients were then assigned to the IST group if they initiated ISTs within the following 7 days, and to the non-IST group otherwise. Importantly, patients were allowed to contribute to multiple trials over time but could only be assigned to the IST group once-at the time they first initiated ISTs. The first day of follow-up (day zero) for each emulated trial was defined as the final day of that trial's enrollment week, and patients were followed until death or the end of the study period (December 31, 2022)
Sampling Method: Non-Probability Sample
Enrollment: 2985 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Relapse | 1 year
  Relapses were identified when patients were treated with one of the following interventions: intravenous steroids, immunoglobulin therapy, or plasma exchange.

SECONDARY OUTCOMES:
Safety outcomes | 6 months after start of ISTs
  Incidence of serious infection, fracture, cancer, myocardial infarction, stroke, depression, anxiety, dementia, and Parkinson's disease which defined as presence of ICD-10 codes.

IPD SHARING:
Plan to Share IPD: No